CLINICAL TRIAL: NCT03397368
Title: Evaluation of Role of Transperineal US in Differentiating Degrees of Genuine Stress Incontinence in Females Diagnosed by Urodynamics
Brief Title: Evaluation of Transperineal US in Stress Incontinence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: stress incontinence
Record Dates: First submitted 2018-01-05; First posted 2018-01-12 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Stress Incontinence, Female
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Urodynamics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transperineal Ultrasound - — Every women with stress incontinence witll be subjected to urodynamics to confirm genuine stress incontinence then will be subjected Transperineal US
  Other Names: Urodynamics

SUMMARY:
Stress urinary incontinence (SUI) has an observed prevalence of between 4%and 35%.Identified risk factors are aging, obesity and repeated pregnancies and deliveries.

Urodynamic remains the gold standard for diagnosis in the past years. Trans labial ultrasound appears to have a good role in diagnosing stress incontinence

DETAILED DESCRIPTION:
A comparative observational cross sectional study will be conducted .

The symptom, or "subjective indicator of disease," of SUI is described as "the complaint of involuntary leakage on effort or exertion, or on sneezing or coughing." 1 Stress urinary incontinence (SUI) has an observed prevalence of between 4% and 35%.

It's a social problem that causes hygienic problem that s distressing for females.

Urodynamic study is the gold standard for diagnosis of most types of urinary incontinence with some limitations as it's not done routinely in all cases of urinary incontinence according to the NICE guidelines 2 Translabial ultrasound is a simple, noninvasive, available, and reproducible method for qualitative and quantitative evaluation of the lower urinary tract in females.

ELIGIBILITY:
Inclusion Criteria:

females between 20-75 years old

* -Women diagnosed to have genuine stress urinary incontinence diagnosed by history taking, voiding diary and confirmed by urodynamic.

Exclusion Criteria:

* -Known to be Diabetic
* Urge incontinence or mixed type
* Voiding dysfunction
* Neurological problems
* open suprapubic wound
* Previous surgery for POP(pelvic organ prolapse) or incontinence
* suspicion of pelvic malignancy

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — females who are complaining from stress incontinence
Study Population: females who are complaining from stress incontinence that did urodynamics study and proved to have a genuine stress incontinence and referred to do transperineal ultrasound
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-11-02 (Estimated); Study Completion 2019-12-08 (Estimated)

PRIMARY OUTCOMES:
The number of participants who will be properly diagnosed to have genuine stress incontinence To determine the role of transperineal ultrasound in diagnosing stress incontinence | within a week
  the outcome describes how much the transperineal us have a power to diagnose stress incontinence in comparison to urodynamic study

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, M.s.c, Study Chair — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (2):
- Egypt (2):
  - Kasralainy Hospital, Cairo
  - Algazeerah, Giza

IPD SHARING:
Plan to Share IPD: No